CLINICAL TRIAL: NCT00286429
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Efficacy and Safety of SYR110322 (SYR-322) When Used in Combination With Insulin in Subjects With Type 2 Diabetes
Brief Title: Efficacy and Safety Study of Alogliptin and Insulin in the Treatment of Type 2 Diabetes.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-322-INS-011; 2005-004671-38 (EudraCT Number); U1111-1113-8369 (Registry Identifier: WHO)
Record Dates: First submitted 2006-02-01; First posted 2006-02-03 (Estimated); Results first posted 2011-08-12 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus; Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Dyslipidemias | interventions — alogliptin; Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin (Placebo Comparator)
  Interventions: Drug: Insulin
- Alogliptin 12.5 mg QD (Experimental)
  Interventions: Drug: Alogliptin and insulin
- Alogliptin 25 mg QD (Experimental)
  Interventions: Drug: Alogliptin and insulin

INTERVENTIONS:
Drug: Alogliptin and insulin — Alogliptin 12.5 mg, tablets, orally, once daily and insulin for up to 26 weeks.
  Other Names: alogliptin; SYR110322
  Arms: Alogliptin 12.5 mg QD
Drug: Alogliptin and insulin — Alogliptin 25 mg, tablets, orally, once daily and insulin for up to 26 weeks.
  Other Names: alogliptin; SYR110322
  Arms: Alogliptin 25 mg QD
Drug: Insulin — Alogliptin placebo-matching tablets, orally, once daily and insulin for up to 26 weeks.
  Arms: Insulin

SUMMARY:
The purpose of this study is to determine the efficacy and safety of alogliptin, once daily (QD), taken in combination with insulin for the treatment of Type 2 Diabetes.

DETAILED DESCRIPTION:
There are approximately 19 million people in the United States who have been diagnosed with diabetes mellitus, of which 90% to 95% are type 2. The prevalence of type 2 diabetes varies among racial and ethnic populations and has been shown to correlate with age, obesity, family history, history of gestational diabetes, and physical inactivity. Over the next decade, a marked increase in the number of adults with diabetes mellitus is expected.

Takeda is developing alogliptin (SYR-322) for patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV enzyme. Dipeptidyl peptidase IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of dipeptidyl peptidase IV will improve glycemic (glucose) control in patients with type 2 diabetes.

The aim of the current study is to evaluate the efficacy of alogliptin in combination with insulin in subjects who are inadequately controlled on insulin alone (with or without metformin). Individuals who participate in this study will be required to commit to a screening visit and up to 14 additional visits at the study center. Study participation is anticipated to be about 34 weeks (or 8.5 months).

ELIGIBILITY:
Inclusion Criteria

* Diagnosis of type 2 diabetes mellitus and currently treated with insulin alone (with or without metformin), and is inadequately controlled. Metformin dose must be stable for at least 8 weeks prior to Randomization.
* No treatment with antidiabetic agents other than insulin and metformin within the 8 weeks prior to Randomization.
* Body mass index greater than or equal to 23 kg/m2 and less than or equal to 45 kg/m2
* Fasting C-peptide concentration greater than or equal to 0.8 ng per mL. (If this screening criterion is not met, the subject still qualifies if C-peptide greater than or equal to 1.5 ng per mL after a challenge test).
* Glycosylated hemoglobin concentration greater than or equal to 8.0% at Screening.
* Using a stable dose of insulin of at least 15 units but not more than 100 units per day for at least 8 weeks prior to Randomization. A dose of insulin that varies by up to 15% of the mean will be considered as stable.
* If regular use of other, non-excluded medications, must be on a stable dose for at least the 4 weeks prior to Screening. However, as needed use of prescription or over-the-counter medications is allowed at the discretion of the investigator.
* Systolic blood pressure less than or equal to180 mm Hg and diastolic pressure less than or equal to 110 mm Hg
* Hemoglobin greater than or equal to 12 g per dL for males and greater than or equal to10 g per dL for females.
* Alanine aminotransferase less than or equal to 3 times the upper limit of normal.
* Serum creatinine less than or equal to 2.0 mg per dL.
* Thyroid-stimulating hormone level less than or equal to the upper limit of the normal range and the subject is clinically euthyroid.
* Neither pregnant (confirmed by laboratory testing in females of childbearing potential) nor lactating.
* Female subjects of childbearing potential must be practicing adequate contraception. Adequate contraception must be practiced for the duration of participation in the study.
* Able and willing to monitor own blood glucose concentrations with a home glucose monitor
* No major illness or debility that in the investigator's opinion prohibits the individual from completing the study
* Able and willing to provide written informed consent

Exclusion Criteria

* Urine albumin to creatinine ratio of greater than 1000 μg per mg at Screening. If elevated, the subject may be rescreened within 1 week.
* History of cancer, other than squamous cell or basal cell carcinoma of the skin, that has not been in full remission for at least 5 years prior to Screening. (History of treated cervical intraepithelial neoplasia I or cervical intraepithelial neoplasia II is allowed.).
* History of laser treatment for proliferative diabetic retinopathy within the 6 months prior to Screening.
* History of treated diabetic gastric paresis.
* New York Heart Association Class III or IV heart failure regardless of therapy. Currently treated subjects who are stable at Class I or II are candidates for the study.
* History of coronary angioplasty, coronary stent placement, coronary bypass surgery, or myocardial infarction within the 6 months prior to Screening.
* History of any hemoglobinopathy that may affect determination of glycosylated hemoglobin.
* History of infection with hepatitis B, hepatitis C, or human immunodeficiency virus.
* History of a psychiatric disorder that will affect ability to participate in the study.
* History of angioedema in association with use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor inhibitors.
* History of alcohol or substance abuse within the 2 years prior to Screening.
* Receipt of any investigational drug within the 30 days prior to Screening or a history of receipt of an investigational antidiabetic drug within the 3 months prior to Screening.
* Prior treatment in an investigational study of alogliptin.
* Excluded Medications:

  * Treatment with antidiabetic agents other than insulin and metformin is not allowed within the 8 weeks prior to Randomization and through the completion of the end-of treatment or early termination procedures. (Exception: if has received other antidiabetic therapy for less than 7 days within the 3 months prior to Screening.)
  * Treatment with weight-loss drugs, any investigational antidiabetics, or oral or systemically injected glucocorticoids is not allowed from 3 months prior to randomization through the completion of the end-of-treatment or early termination procedures. Inhaled corticosteroids are allowed.
  * Must not take any medications, including over-the-counter products, without first consulting with the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2006-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda
Locations (60):
- United States (45):
  - Phoenix, Arizona
  - Anaheim, California
  - Artesia, California
  - Fresno, California
  - Mission Viejo, California
  - Northridge, California
  - Orange, California
  - San Diego, California
  - Tustin, California
  - Walnut Creek, California
  - Denver, Colorado
  - Cocoa Beach, Florida
  - Longwood, Florida
  - New Port Richey, Florida
  - Ocala, Florida
  - Saint Cloud, Florida
  - Tampa, Florida
  - Lawrenceville, Georgia
  - Honolulu, Hawaii
  - Avon, Indiana
  - Evansville, Indiana
  - Lafayette, Indiana
  - St Louis, Missouri
  - Omaha, Nebraska
  - Berlin, New Jersey
  - Burlington, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Morehead City, North Carolina
  - Pinehurst, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Tulsa, Oklahoma
  - Medford, Oregon
  - Lansdale, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Simpsonville, South Carolina
  - Cookeville, Tennessee
  - Corpus Christi, Texas
  - Dallas, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Texarkana, Texas
  - Burlington, Vermont
- Multiple Cities, Argentina
- Multiple Cities, Australia
- Multiple Cities, Brazil
- Multiple Cities, Chile
- Multiple Cities, Czechia
- Multiple Cities, Germany
- Multiple Cities, Guatemala
- Multiple Cities, Hungary
- Multiple Cities, India
- Multiple Cities, Mexico
- Multiple Cities, Netherlands
- Multiple Cities, New Zealand
- Multiple Cities, Peru
- Multiple Cities, Poland
- Multiple Cities, South Africa

REFERENCES:
- [Result] Rosenstock J, Rendell MS, Gross JL, Fleck PR, Wilson CA, Mekki Q. Alogliptin added to insulin therapy in patients with type 2 diabetes reduces HbA(1C) without causing weight gain or increased hypoglycaemia. Diabetes Obes Metab. 2009 Dec;11(12):1145-52. doi: 10.1111/j.1463-1326.2009.01124.x. Epub 2009 Sep 16. PMID 19758359
- [Result] Pratley RE, McCall T, Fleck PR, Wilson CA, Mekki Q. Alogliptin use in elderly people: a pooled analysis from phase 2 and 3 studies. J Am Geriatr Soc. 2009 Nov;57(11):2011-9. doi: 10.1111/j.1532-5415.2009.02484.x. Epub 2009 Sep 30. PMID 19793357

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 110 investigative sites in Australia, Brazil, Chile, Guatemala, Germany, Hungary, India, Mexico, New Zealand, the Netherlands, Poland, South Africa, and the United States from 16 March 2006 to 18 September 2006
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus who were inadequately controlled while being treated with insulin with or without metformin were enrolled in one of three, once-daily (QD) treatment groups.
Groups:
- Placebo: Alogliptin placebo-matching tablets, orally, once daily and insulin for up to 26 weeks.
- Alogliptin 12.5 mg QD: Alogliptin 12.5 mg, tablets, orally, once daily and insulin for up to 26 weeks.
- Alogliptin 25 mg QD: Alogliptin 25 mg, tablets, orally, once daily and insulin for up to 26 weeks.
Period: Overall Study
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Started | 130 | 131 | 129
Completed | 55 | 83 | 77
Not Completed | 75 | 48 | 52
Not completed — Adverse Event | 4 | 1 | 6
Not completed — Lack of Efficacy | 52 | 27 | 25
Not completed — Lost to Follow-up | 2 | 4 | 3
Not completed — Physician Decision | 10 | 7 | 7
Not completed — Protocol Violation | 3 | 5 | 4
Not completed — Withdrawal by Subject | 3 | 2 | 6
Not completed — Administrative Error | 1 | 1 | 1
Not completed — Administrative Decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD | Total
Number analyzed (Participants) | 130 | 131 | 129 | 390
Age, Customized [Number; unit: participants]
  <65 years | 109 | 112 | 106 | 327
  ≥65 years | 21 | 19 | 23 | 63
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 76 | 85 | 229
  Male | 62 | 55 | 44 | 161

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Glycosylated Hemoglobin (HbA1c) at Week 26.
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 26 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF). ANCOVA = Analysis of covariance.
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 126 | 130 | 126
percentage of Glycosylated Hemoglobin | -0.13 (0.077) | -0.63 (0.076) | -0.71 (0.078)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c at Week 26. For comparison of either alogliptin dose vs. placebo (2-sample t test), study sample size >=390 participants had 95% power to detect a treatment difference as small as 0.4% in the per protocol analysis set assuming a standard deviation of 0.8%, a 2-sided test at 0.05 significance level and >=80% of subjects meeting the per protocol criteria; Test type: Superiority or Other; p < 0.001, ANCOVA — A step-down strategy was used for the primary analysis. First, the 25mg dose was compared to placebo at the 2-sided 0.05 significance level. The 12.5 mg dose was compared to placebo only if the comparison of the 25mg dose to placebo was significant; ANCOVA included treatment, geographic region, and baseline metformin regimen as class variables, and baseline covariates (insulin dose and HbA1c); Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.72 to -0.30] — Negative mean treatment difference indicates larger decrease from baseline (more negative change from baseline) in the alogliptin arm compared to the placebo arm
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.80 to -0.37] — [estimate comment as in outcome 1, analysis 1]

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 4).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 4 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized participants who received at least 1 dose of study drug and who had an HbA1c measurement at baseline and at Week 4. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 114 | 116 | 116
percentage of Glycosylated Hemoglobin | -0.26 (0.045) | -0.47 (0.045) | -0.58 (0.045)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c at Week 4. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.34 to -0.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.32, 95% CI 2-sided [-0.45 to -0.20] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 8. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 126 | 130 | 126
percentage of Glycosylated Hemoglobin | -0.27 (0.061) | -0.76 (0.060) | -0.84 (0.062)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c at Week 8. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.48, 95% CI 2-sided [-0.65 to -0.31] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.56, 95% CI 2-sided [-0.73 to -0.39] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 12. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 126 | 130 | 126
percentage of Glycosylated Hemoglobin | -0.27 (0.073) | -0.84 (0.072) | -0.81 (0.073)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c at Week 12. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.77 to -0.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.75 to -0.34] — [estimate comment as in outcome 1, analysis 1]

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 16. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 126 | 130 | 126
percentage of Glycosylated Hemoglobin | -0.22 (0.076) | -0.80 (0.074) | -0.76 (0.076)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c at Week 16. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.79 to -0.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.54, 95% CI 2-sided [-0.75 to -0.33] — [estimate comment as in outcome 1, analysis 1]

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of Glycosylated Hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and Glycosylated Hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 20. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 126 | 130 | 126
percentage of Glycosylated Hemoglobin | -0.17 (0.078) | -0.76 (0.076) | -0.74 (0.078)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in HbA1c at Week 20. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.80 to -0.37] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.79 to -0.35] — [estimate comment as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 1).
Description: The change between the value of fasting plasma glucose collected at final visit or week 1 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 1.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 1. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 107 | 121 | 111
mg/dL | 6.3 (5.40) | -5.0 (5.07) | -9.9 (5.33)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 1. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.128, ANCOVA — No multiplicity adjustments; ANCOVA included treatment, geographic region, and baseline metformin regimen as class variables, and baseline covariates (insulin dose and FPG); Mean Difference (Final Values) = -11.3, 95% CI 2-sided [-25.9 to 3.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 7, analysis 1]; Test type: Superiority or Other; p = 0.034, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -16.1, 95% CI 2-sided [-31.1 to -1.2] — [estimate comment as in outcome 1, analysis 1]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 2).
Description: The change between the value of fasting plasma glucose collected at week 2 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 2.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 2. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 115 | 127 | 119
mg/dL | 1.0 (5.09) | -3.1 (4.84) | -11.4 (5.03)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 25 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 2. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.563, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -4.1, 95% CI 2-sided [-17.9 to 9.7] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 8, analysis 1]; Test type: Superiority or Other; p = 0.084, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -12.4, 95% CI 2-sided [-26.4 to 1.7] — [estimate comment as in outcome 1, analysis 1]

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 4).
Description: The change between the value of fasting plasma glucose collected at week 4 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 4.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 4. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 119 | 128 | 120
mg/dL | 5.3 (5.28) | -5.0 (5.08) | -12.1 (5.28)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 4. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.160, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -10.3, 95% CI 2-sided [-24.7 to 4.1] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 9, analysis 1]; Test type: Superiority or Other; p = 0.020, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -17.4, 95% CI 2-sided [-32.1 to -2.8] — [estimate comment as in outcome 1, analysis 1]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 124 | 131 | 126
mg/dL | 5.4 (5.42) | -13.5 (5.26) | -14.1 (5.39)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 8. The treatment effect was be evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.013, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -18.9, 95% CI 2-sided [-33.7 to -4.0] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 8. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.011, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -19.5, 95% CI 2-sided [-34.5 to -4.5] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 127 | 131 | 128
mg/dL | -1.4 (5.47) | -5.2 (5.38) | -2.9 (5.47)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 12. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.624, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -3.8, 95% CI 2-sided [-18.9 to 11.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 11, analysis 1]; Test type: Superiority or Other; p = 0.853, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-16.7 to 13.8] — [estimate comment as in outcome 1, analysis 1]

12. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 16).
Description: The change between the value of fasting plasma glucose collected at week 16 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 127 | 131 | 128
mg/dL | 4.6 (5.38) | -5.3 (5.29) | -6.3 (5.38)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 16. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.190, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -9.9, 95% CI 2-sided [-24.7 to 4.9] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 16. The treatment effect was be evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.154, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -10.9, 95% CI 2-sided [-25.8 to 4.1] — [estimate comment as in outcome 1, analysis 1]

13. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 20).
Description: The change between the value of fasting plasma glucose collected at week 20 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 127 | 131 | 128
mg/dL | 8.6 (5.45) | -4.2 (5.36) | -11.3 (5.46)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 20. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.097, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -12.7, 95% CI 2-sided [-27.8 to 2.3] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 13, analysis 1]; Test type: Superiority or Other; p = 0.010, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -19.9, 95% CI 2-sided [-35.1 to -4.7] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 26).
Description: The change between the value of fasting plasma glucose collected at week 26 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 26.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had measurements at baseline and at Week 26. Missing data are imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 127 | 131 | 128
mg/dL | 5.8 (5.69) | 2.3 (5.59) | -11.7 (5.69)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in FPG at Week 26. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.662, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -3.5, 95% CI 2-sided [-19.2 to 12.2] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 14, analysis 1]; Test type: Superiority or Other; p = 0.030, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 7, analysis 1]; Mean Difference (Final Values) = -17.6, 95% CI 2-sided [-33.4 to -1.7] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Number of Participants With Marked Hyperglycemia (Fasting Plasma Glucose ≥ 200 mg Per dL).
Description: The number of participants with a fasting plasma glucose value greater than or equal to 200 mg per dL during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had at least 1 fasting plasma glucose measurement after baseline.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 128 | 131 | 128
participants | 105 | 99 | 86
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in number of participants with marked hyperglycemia. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p = 0.075, Regression, Logistic — No multiplicity adjustments; Logistic regression model includes effects for treatment, geographic region, baseline metformin regimen, baseline insulin dose, and baseline HbA1c; Odds Ratio (OR) = 0.551, 95% CI 2-sided [0.286 to 1.063] — Odds Ratio (OR) is alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 15, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 0.364, 95% CI 2-sided [0.191 to 0.695] — Odds Ratio (OR) is alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

16. Secondary Outcome: Number of Participants Requiring Rescue.
Description: The number of participants requiring rescue for failing to achieve pre-specified glycemic targets during the 26 week study.
Time Frame: 26 Weeks.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who completed at least 1 study visit after baseline.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 128
participants | 52 | 27 | 25
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in number of participants requiring rescue. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 0.350, 95% CI 2-sided [0.198 to 0.619] — Odds Ratio (OR) is alogliptin arm versus placebo arm. OR <1.0 indicates lower incidence compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 16, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 0.339, 95% CI 2-sided [0.189 to 0.608] — Odds Ratio (OR) is alogliptin arm versus placebo. OR <1.0 indicates lower incidence compared to placebo

17. Secondary Outcome: Change From Baseline in C-peptide (Week 4).
Description: The change between the value of C-peptide collected at week 4 and C-peptide collected at baseline.
Time Frame: Baseline and Week 4.
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 99 | 111 | 109
ng/mL | -0.023 (0.1062) | 0.132 (0.1001) | 0.453 (0.1014)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in C-Peptide at Week 4. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.286, ANCOVA — No multiplicity adjustments; ANCOVA included treatment, geographic region, and baseline metformin regimen as class variables, and baseline covariates (insulin dose and C-peptide); Mean Difference (Final Values) = 0.156, 95% CI 2-sided [-0.131 to 0.443] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 17, analysis 1]; Test type: Superiority or Other; p = 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = .477, 95% CI 2-sided [0.188 to 0.765] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Change From Baseline in C-peptide (Week 8).
Description: The change between the value of C-peptide collected at week 8 and C-peptide collected at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 121 | 130 | 123
ng/mL | -0.024 (0.1224) | 0.178 (0.1180) | 0.348 (0.1220)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in C-Peptide at Week 8. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.236, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.202, 95% CI 2-sided [-0.132 to 0.536] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 18, analysis 1]; Test type: Superiority or Other; p = 0.032, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.372, 95% CI 2-sided [0.032 to 0.712] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Change From Baseline in C-peptide (Week 12).
Description: The change between the value of C-peptide collected at week 12 and C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 124 | 130 | 126
ng/mL | 0.207 (0.1558) | 0.333 (0.1521) | 0.390 (0.1553)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in C-peptide at Week 12. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.562, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.126, 95% CI 2-sided [-0.302 to 0.554] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 19, analysis 1]; Test type: Superiority or Other; p = 0.407, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.183, 95% CI 2-sided [-0.251 to 0.616] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Change From Baseline in C-peptide (Week 16).
Description: The change between the value of C-peptide collected at week 16 and C-peptide collected at baseline.
Time Frame: Baseline and Week 16.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 124 | 130 | 126
ng/mL | 0.241 (0.1536) | 0.319 (0.1500) | 0.396 (0.1532)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in C-peptide at Week 16. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.716, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [-0.344 to 0.500] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 20, analysis 1]; Test type: Superiority or Other; p = 0.474, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.156, 95% CI 2-sided [-0.272 to 0.583] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Change From Baseline in C-peptide (Week 20).
Description: The change between the value of C-peptide collected at week 20 and C-peptide collected at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 124 | 130 | 126
ng/mL | 0.239 (0.1467) | 0.318 (0.1432) | 0.281 (0.1463)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in C-peptide at Week 20. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.700, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.079, 95% CI 2-sided [-0.324 to 0.482] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 21, analysis 1]; Test type: Superiority or Other; p = 0.839, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.042, 95% CI 2-sided [-0.366 to 0.450] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Change From Baseline in C-peptide (Week 26).
Description: The change between the value of C-peptide collected at week 26 or final visit and C-peptide collected at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: ng/mL
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 124 | 130 | 126
ng/mL | -0.083 (0.1192) | 0.199 (0.1164) | 0.042 (0.1189)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in C-peptide at Week 26. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.091, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.282, 95% CI 2-sided [-0.045 to 0.610] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 22, analysis 1]; Test type: Superiority or Other; p = 0.459, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = 0.125, 95% CI 2-sided [-0.207 to 0.457] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 6.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 6.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who completed at least 1 HbA1c measurement after baseline.
  Due to no participants in the placebo arm achieved HbA1c ≤ 6.5%, the odds ratio of alogliptin to placebo and 95% CI were not estimable from the logistic regression.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 129
participants | 0 | 3 | 3

24. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.0%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 7.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had at least 1 HbA1c measurement after baseline.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 129
participants | 1 | 11 | 10
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in incidence of HbA1c ≤7.0%. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p = 0.016, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 12.650, 95% CI 2-sided [1.589 to 100.682] — Odds Ratio (OR) compares alogliptin arm versus placebo. OR >1.0 indicates higher incidence of response compared to placebo
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in incidence of HbA1c ≤7.0%. The treatment effect was evaluated as a contrast of each active dose versus placebo was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p = 0.023, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 11.255, 95% CI 2-sided [1.401 to 90.379] — [estimate comment as in outcome 24, analysis 1]

25. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin ≤ 7.5%.
Description: The number of participants with a value for the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) less than or equal to 7.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 129
participants | 5 | 22 | 33
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in incidence of HbA1c ≤7.5%. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 5.777, 95% CI 2-sided [2.047 to 16.305] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 25, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 9.784, 95% CI 2-sided [3.540 to 27.039] — [estimate comment as in outcome 24, analysis 1]

26. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 0.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 0.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 129
participants | 40 | 70 | 70
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in incidence of HbA1c decrease from baseline ≥0.5%. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 2.674, 95% CI 2-sided [1.579 to 4.530] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 26, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 2.819, 95% CI 2-sided [1.653 to 4.808] — [estimate comment as in outcome 24, analysis 1]

27. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 129
participants | 17 | 41 | 47
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD vs Alogliptin 25 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in incidence of HbA1c decrease from baseline ≥1.0%. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 3.163, 95% CI 2-sided [1.651 to 6.060] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 27, analysis 1]; Test type: Superiority or Other; p < 0.001, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 3.989, 95% CI 2-sided [2.083 to 7.640] — [estimate comment as in outcome 24, analysis 1]

28. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 1.5%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 1.5% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: as for outcome 24
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 129
participants | 6 | 22 | 23
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no treatment effect between alogliptin and placebo arms in incidence of HbA1c decrease from baseline ≥1.5%. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a Wald test at the 0.05 significance level; Test type: Superiority or Other; p = 0.002, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 4.550, 95% CI 2-sided [1.732 to 11.953] — [estimate comment as in outcome 24, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 28, analysis 1]; Test type: Superiority or Other; p = 0.002, Regression, Logistic — No multiplicity adjustments; [statistical method as in outcome 15, analysis 1]; Odds Ratio (OR) = 4.580, 95% CI 2-sided [1.740 to 12.052] — [estimate comment as in outcome 24, analysis 1]

29. Secondary Outcome: Number of Participants With Glycosylated Hemoglobin Decrease From Baseline ≥ 2.0%.
Description: The number of participants with a decrease from baseline in the percentage of glycosylated hemoglobin (the percentage of hemoglobin that is bound to glucose) greater than or equal to 2.0% during the 26 week study.
Time Frame: Baseline and Week 26.
Population: Randomized subjects who received at least 1 dose of study drug (Full Analysis Set), and who had at least 1 HbA1c measurement after baseline.
  Due to no participants in the placebo arm achieved HbA1c decrease from baseline ≥2.0%, the odds ratio of alogliptin to placebo and 95% CI were not estimable from the logistic regression.
Measure: Number; unit: participants
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 129 | 131 | 129
participants | 0 | 11 | 11

30. Secondary Outcome: Change From Baseline in Body Weight (Week 8).
Description: The change between Body Weight measured at week 8 and Body Weight measured at baseline.
Time Frame: Baseline and Week 8.
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 118 | 125 | 121
kg | 0.39 (0.191) | 0.10 (0.185) | 0.18 (0.189)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in body weight at Week 8. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.291, ANCOVA — No multiplicity adjustments; ANCOVA included treatment, geographic region, and baseline metformin regimen as class variables, and baseline covariates (insulin dose and weight); Mean Difference (Final Values) = -0.28, 95% CI 2-sided [-0.81 to 0.24] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 30, analysis 1]; Test type: Superiority or Other; p = 0.439, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.21, 95% CI 2-sided [-0.74 to 0.32] — [estimate comment as in outcome 1, analysis 1]

31. Secondary Outcome: Change From Baseline in Body Weight (Week 12).
Description: The change between Body Weight measured at week 12 and Body Weight measured at baseline.
Time Frame: Baseline and Week 12.
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 121 | 127 | 123
kg | 0.50 (0.221) | 0.44 (0.215) | 0.31 (0.219)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in body weight at Week 12. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.841, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.67 to 0.55] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 31, analysis 1]; Test type: Superiority or Other; p = 0.556, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.80 to 0.43] — [estimate comment as in outcome 1, analysis 1]

32. Secondary Outcome: Change From Baseline in Body Weight (Week 20).
Description: The change between Body Weight measured at week 20 and Body Weight measured at baseline.
Time Frame: Baseline and Week 20.
Population: as for outcome 6
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 121 | 127 | 124
kg | 0.73 (0.231) | 0.55 (0.225) | 0.45 (0.229)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in body weight at Week 20. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.586, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.81 to 0.46] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 32, analysis 1]; Test type: Superiority or Other; p = 0.404, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.27, 95% CI 2-sided [-0.91 to 0.37] — [estimate comment as in outcome 1, analysis 1]

33. Secondary Outcome: Change From Baseline in Body Weight (Week 26).
Description: The change between Body Weight measured at week 26 or final visit and Body Weight measured at baseline.
Time Frame: Baseline and Week 26.
Population: as for outcome 14
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Number analyzed (Participants) | 121 | 127 | 124
kg | 0.63 (0.244) | 0.68 (0.237) | 0.60 (0.241)
Statistical Analysis 1: Comparison: Placebo vs Alogliptin 12.5 mg QD; The null hypothesis that there is no difference between alogliptin and placebo arms in change from baseline in body weight at Week 26. The treatment effect was evaluated as a contrast of each active dose versus placebo and was evaluated inferentially with a 2-sided t test at the 0.05 significance level; Test type: Superiority or Other; p = 0.874, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = 0.05, 95% CI 2-sided [-0.62 to 0.72] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Alogliptin 25 mg QD; [analysis description as in outcome 33, analysis 1]; Test type: Superiority or Other; p = 0.948, ANCOVA — No multiplicity adjustments; [statistical method as in outcome 30, analysis 1]; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.70 to 0.65] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of double-blind study drug and no more than 14 days (or 30 days for a serious event) after the last dose of double-blind drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was was recorded, irrespective of the relation to study treatment.
Arm/Group | Placebo | Alogliptin 12.5 mg QD | Alogliptin 25 mg QD
Serious Adverse Events (participants affected / at risk) | 6/129 | 8/131 | 7/129
Other Adverse Events (participants affected / at risk) | 54/129 | 58/131 | 50/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=129) | Alogliptin 12.5 mg QD (N=131) | Alogliptin 25 mg QD (N=129)
Angina unstable (Cardiac disorders) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Demyelination (Nervous system disorders) | 1 | 0 | 0
Diverticulitis intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Hypoglycaemic coma (Nervous system disorders) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1 | 0
Scrotal abscess (Infections and infestations) | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 1
Sudden death (General disorders) | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=129) | Alogliptin 12.5 mg QD (N=131) | Alogliptin 25 mg QD (N=129)
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 9 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 2 | 6
Bronchitis (Infections and infestations) | 4 | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 7 | 1 | 8
Dizziness (Nervous system disorders) | 2 | 5 | 1
Headache (Nervous system disorders) | 6 | 7 | 4
Hypertension (Vascular disorders) | 6 | 5 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 3 | 5 | 2
Influenza (Infections and infestations) | 3 | 4 | 3
Insomnia (Psychiatric disorders) | 0 | 4 | 1
Nasopharyngitis (Infections and infestations) | 6 | 5 | 8
Nausea (Gastrointestinal disorders) | 3 | 4 | 6
Oedema peripheral (General disorders) | 4 | 4 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 4
Upper respiratory tract (Infections and infestations) | 4 | 6 | 4
Urinary tract infection (Infections and infestations) | 10 | 8 | 9
Vomiting (Gastrointestinal disorders) | 4 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication related to study results will be published prior to publication of a multi-center report submitted for publication within 18 months after conclusion or termination of a study at all study sites. Results publications will be submitted to sponsor for review 60 days in advance of publication. Sponsor can require removal of confidential information unrelated to study results. Sponsor can embargo a proposed publication for another 60 days to preserve intellectual property.